CLINICAL TRIAL: NCT03065322
Title: The Impact of Obstructive Sleep Apnoea in Women With Polycystic Ovary Syndrome: A Cross-sectional Study
Brief Title: The Impact of Obstructive Sleep Apnoea in Women With Polycystic Ovary Syndrome.
Status: Completed | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: University of Warwick (Other)
Responsible Party: Sponsor
Other Study IDs: MW181216; 213996 (Other: IRAS)
Record Dates: First submitted 2017-01-12; First posted 2017-02-27 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Polycystic Ovary Syndrome; Obstructive Sleep Apnea
Keywords: PCOS; OSA
MeSH Terms: conditions — Polycystic Ovary Syndrome; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with PCOS: Women with confirmed diagnosis of PCOS, based on the Rotterdam Criteria. To assess risk of OSA: the risk of OSA will be assessed using the Berlin questionnaire and the Epworth Sleepiness Scale (ESS). Women with at high risk of OSA will have home-based sleep studies performed.
  Interventions: Other: To assess risk of OSA

INTERVENTIONS:
Other: To assess risk of OSA — The risk of OSA will be assessed using the Berlin questionnaire and the Epworth Sleepiness Scale (ESS). Women with at high risk of OSA will have home-based sleep studies performed. Study participants will be divided based on the results of the Berlin and ESS questionnaires and sleep studies into two groups: 1) PCOS low risk OSA: women with normal ESS and normal Berlin questionnaire (no sleep studies performed), or women with normal sleep studies; and 2) PCOS OSA: women with OSA proven by sleep studies.

SUMMARY:
Women with PCOS and OSA, compared to women with PCOS only, have more severe clinical and biochemical features of PCOS and impaired QoL. This is an observational cross-sectional study in a secondary care PCOS clinic in the WISDEM Centre, University Hospital Coventry.

The primary aim of this study is to examine the relationship between OSA and impaired QoL in women with PCOS. Study secondary outcomes are to examine the relationship between OSA and the clinical and biochemical features in women with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in women of reproductive age. PCOS is associated with multiple co-morbidities including obesity, insulin resistance, subfertility, impaired quality of life (QoL) and increased risk of type 2 diabetes. Obstructive sleep apnoea (OSA) is a common medical condition that is often undiagnosed, particularly in women. Obesity is a common risk factor for OSA and PCOS and OSA is associated with comorbidities similar to those observed in patients with PCOS such as insulin resistance, increased risk of type 2 diabetes, and impaired QoL. Hence it is not surprising that OSA and PCOS might co-exist.

However, the impact of OSA in women with PCOS remains unclear and understudied. It is plausible that OSA may contribute to the subfertility and impaired QoL observed in women with PCOS by increasing insulin resistance, activation of the sympathetic nervous system, disturbing the hypothalamic/pituitary/ovarian axis, and contributing to excessive daytime sleepiness and reduced mood.

38 women with PCOS will be recruited from the PCOS clinic, weight management clinic, reproductive endocrinology clinic and through posters displayed at University Hospital Coventry and an e-poster displayed at the hospital intranet. Women with increased risk of OSA, based on the Berlin questionnaire and the Epworth Sleepiness Scale (ESS), will have home-based sleep studies performed. They will also be referred to the Respiratory Physician, as part of routine NHS care.

Study participants will be divided based on the results of the Berlin and ESS questionnaires and sleep studies into two groups: 1) PCOS low risk OSA: women with normal ESS and normal Berlin questionnaire (no sleep studies performed), or women with normal sleep studies; and 2) PCOS OSA: women with OSA proven by sleep studies.

Clinical and biochemical features including reproductive history, depression and anxiety [using the Hospital Anxiety and Depression questionnaire (HAD)], and QoL [using the PCOS health-related quality of life questionnaire (PCOSQ) and the World Health Organisation QoL-BREF will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS, defined by the Rotterdam criteria as 2 out of 3:

  1. Oligo/anovulation 2. Clinical or biochemical evidence of hirsutism 3. Polycystic ovaries on ultrasound. And the exclusion of other disorders with similar presentation including: non-classic congenital adrenal hyperplasia, androgen secreting tumours, Cushing's syndrome; thyroid disorders and prolactinomas.
* Age ≥ 18 years.
* Able to provide written consent.
* Able to adequately understand English.
* Patients with unknown diagnosis of OSA, or who were investigated in the past and either found not to have OSA, or found to have OSA and are not on CPAP therapy.

Exclusion Criteria:

* Pregnancy or breastfeeding women.
* Patients who are unable to give consent.
* Patients known to have OSA treated with CPAP.
* Anyone under the age of 18 years.
* Unable to adequately understand or speak English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with PCOS will be recruited consecutively from the PCOS clinic at the WISDEM centre, University Hospital Coventry. In addition, patient information sheet (PIS) and a study invitation letter will be sent to women with PCOS who attended the PCOS clinic in the last 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Difference in scores on the World Health Organisation QoL questionnaire (WHOQOL-BREF) between women with PCOS and low risk of OSA compared to women with PCOS and OSA. | One day.
  Quality of life will be measured using the World Health Organisation QoL-BREF (WHOQOL-BREF) questionnaire.

SECONDARY OUTCOMES:
Difference in BMI between women with PCOS and low risk of OSA compared to women with PCOS and OSA. | One day.
  BMI will be calculated as kg/m2
Difference in the number of periods per year between women with PCOS and low risk of OSA compared to women with PCOS and OSA | One day.
  Participants will be asked to recall how many periods they had in the last 4 months.
Difference in scores on the Hospital Anxiety and Depression (HAD) scale between women with PCOS and low risk of OSA compared to women with PCOS and OSA. | One day.
  Participants will be asked to complete HAD questionnaire.
Difference in the levels of HOMA-IR between women with PCOS and low risk of OSA compared to women with PCOS and OSA in women with PCOS. | One day.
  Fasting plasma glucose and insulin will be measured to calculate HOMA-IR
Difference in scores on the PCOS health-related quality of life questionnaire (PCOSQ) between women with PCOS and low risk of OSA compared to women with PCOS and OSA. | One day
  Quality of life will be measured using the PCOS health-related quality of life questionnaire (PCOSQ).
Difference in modified Ferriman-Gallwey score between women with PCOS and low risk of OSA compared to women with PCOS and OSA. | One day.
  Hirsutism will be measured using the modified Ferriman-Gallwey score.
Difference in the levels of testosterone between women with PCOS and low risk of OSA compared to women with PCOS and OSA in women with PCOS. | One day.
  Testosterone will be measured in nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Martin O Weickert, MD, FRCP, Principal Investigator — University Hospitals Coventry and Warwickshire NHS Trust
Locations (1):
- University Hospitals Coventry & Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom

REFERENCES:
- [Derived] Kahal H, Tahrani AA, Kyrou I, Dimitriadis GK, Kimani PK, Barber TM, Nicholls M, Ali A, Weickert MO, Randeva HS. The relationship between obstructive sleep apnoea and quality of life in women with polycystic ovary syndrome: a cross-sectional study. Ther Adv Endocrinol Metab. 2020 Feb 21;11:2042018820906689. doi: 10.1177/2042018820906689. eCollection 2020. PMID 32128106

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT03065322/Prot_SAP_000.pdf